CLINICAL TRIAL: NCT00752817
Title: Creating and Implementing a Proficiency-Based Progression Virtual Reality Training Programme for Higher Surgical Trainees for Laparoscopic Assisted Sigmoid Colectomy.
Brief Title: Creating a Proficiency-Based Virtual Reality Simulation Training Programme for Laparoscopic Assisted Colectomy
Acronym: LAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Health Service Executive (Unknown)
Responsible Party: Professor Anthony Gallagher, PhD, Royal College of Surgeons in Ireland (RCSI)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: RCSI 3
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Colorectal Disease
Keywords: Virtual Reality; Simulator; Proficiency; Laparoscopic; Colectomy; Education; Surgical Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SC (Experimental): Subjects (surgical trainees) randomised to train under a proficiency-based progression virtual reality simulation curriculum
  Interventions: Other: Proficiency-based virtual reality simulation training
- CC (Active Comparator): Subjects (surgical trainees) randomised to the current surgical training curriculum
  Interventions: Other: Training under the current surgical training programme

INTERVENTIONS:
Other: Proficiency-based virtual reality simulation training — Subjects (surgical trainees) will be trained under a proficiency-based virtual reality simulation training programme before performing their first live case
  Other Names: Simulation Curriculum; SC
  Arms: SC
Other: Training under the current surgical training programme — Subjects (surgical trainees) will continue to train under the current training methodology offered at their institution before they perform their first live case.
  Other Names: Current Curriculum; CC
  Arms: CC

SUMMARY:
Laparoscopic Colectomy is an advanced minimally invasive procedure that requires advanced laparoscopic skills.

Minimally invasive surgery offers many advantages to the patients but exposes the surgeon to new challenges, many of which are human factor in nature. This in turn prolongs the learning curve and has delayed the widespread adoption of minimally invasive surgical techniques in the management of patients with colorectal disease.

Virtual reality simulation offers an effective way of training whereby surgical trainees can train repeatedly and achieve proficiency in a shorter time and a safe environment.

DETAILED DESCRIPTION:
Introduction:

Minimally Invasive Surgery (MIS) has conferred considerable advantages on patient's post operative outcome and recovery when compared with open surgery.

Major clinical trials including; Clinical Outcomes of Surgical Therapy Study Group (COSTSG), Colon Cancer Laparoscopic or Open Resection (COLOR), and Conventional vs. Laparoscopic-Assisted Surgery in Colorectal Cancer (CLASICC) have uniformly and consistently shown a significant reduction in the post operative pain, the use of narcotics and oral analgesics, and length of hospital stay, as well as a faster resumption of diet, return of bowel function when using a MIS approach.

Despite all these advantages to the patients, MIS imposed a significant difficulty on the surgeons. These difficulties were primarily human factor in nature.

The use of Virtual Reality (VR) simulation has been proven to help in the acquisition of MIS skills. The use of proficiency-based, virtual reality simulation should help training of MIS providers in a safe environment where complex tasks can be repeated as many times as needed to achieve a pre-set proficiency level. A well designed proficiency-based simulation curriculum should help the widespread use of the MIS approach.

Aims

Primary:

We aim to prove that subjects randomised to train under a proficiency-based progression simulation curriculum (SC) will learn to perform laparoscopic assisted colectomy faster, complete more surgical steps and commit fewer operative errors compared to subjects randomised to the current surgical training curriculum (CC)

Secondary:

We aim to set the institutional and national proficiency level for Laparoscopic Assisted Colectomy (LAC) using the ProMIS-LAC simulator from Haptica, Ireland.

Methods Randomised, controlled, single blinded, multicentre study. Primary Variable 8 centres, 8 co-investigators (expert consultant laparoscopic colorectal surgeons > 300 MIS procedures) and 16 surgical trainees will be recruited for the study. Subjects (surgical trainees) will be randomised into;

* Simulator Curriculum (SC) group.
* Conventional Curriculum (CC) group.

Subjects randomised to the CC group will continue to have the conventional training programme offered at their respective hospitals. Subjects randomised to the SC group will complete a standardised laparoscopic skills training course followed by a training curriculum including the performance of simulated LAC procedures in nine predetermined steps on the simulator. Subjects must reach a predetermined proficiency level to complete the simulation training course before re-joining their training programme offered at their respective hospitals. .

Upon completion of the training courses, both groups' subject populations will perform a total of five LAC procedures on consecutive patients in the presence of a surgeon proctor.

Patients indicated for LAC procedure will be screened, consented, and enrolled as patients into this study. Each procedure will be recorded and forwarded to the chief investigator for analysis. The number of completed surgical steps and the incidence of intraoperative errors between the two SC and CC groups will be evaluated via blinded video review.

Secondary Variable

All participating co-investigators will participate in defining the proficiency level for LAC on the ProMIS-LAC simulator.

The average values of the recorded metrics which are obtained from the expert performance will be used to set the proficiency level.

ELIGIBILITY:
Inclusion criteria for subjects

* Classified as year 3-5 post graduation registrars, specialist registrars or residents in surgery.
* Completed their Basic Surgical Training programme.
* Completed at least 12 months period on a Higher Surgical Training programme.
* In an accredited surgical post at time of participation
* In a colorectal surgery rotation at time of participation
* Signed their own consent form

Exclusion criteria for subjects

* Performed, as primary surgeon, > 10 advanced laparoscopic procedures (laparoscopic cholecystectomy, inguinal hernia, appendectomy, Nissen fundoplication, or ventral incisional hernia repair are not considered advanced laparoscopic procedures )
* Performed, as primary surgeon, laparoscopic assisted colectomy procedures
* Performed, as primary surgeon, any hand-assisted laparoscopic colectomy procedures
* Did not sign their own consent form

Inclusion criteria for patients

* Indicated for a laparoscopic assisted sigmoid colectomy or high anterior resection
* At least 18 years old upon date of signing the informed consent document (ICD)
* Sign their own ICD

Exclusion criteria for patients

* History or current diagnosis of synchronous colon cancer
* Indicated for urgent surgery
* Indicated for diverting stoma
* American Society of Anaesthesiologists (ASA) Classification of Physical Status IV-V
* Tumour classified as T4
* An obstructed colon
* Planned early conversion based on findings at operative visualisation.
* Pregnancy
* < 18 years of age
* Mental disability
* Did not sign their own ICD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Subjects randomised to train under a proficiency-based simulation curriculum (SC) will perform laparoscopic assisted colectomy faster, complete more surgical steps and commit fewer operative errors compared to subjects randomised to the control group | 6-12 months

SECONDARY OUTCOMES:
We aim to set the institutional and national proficiency level for Laparoscopic Assisted Colectomy (LAC) using the ProMIS-LAC simulator from Haptica, Ireland. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul Neary, MD, FRCSI, Principal Investigator — Royal College of Surgeons in Ireland
Locations (9):
- Ireland (5):
  - Mercy University Hospital, Cork
  - AMNCH, Dublin
  - St. Vincent's University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Tullamore general hospital, Tullamore
- United Kingdom (4):
  - Antrim Area Hospital, Antrim
  - Gartnavel General Hospital, Glasgow
  - Leicester Royal Infirmary Hospital, Leicester
  - Freeman Hospital, Newcastle

REFERENCES:
- [Background] Ahlberg G, Enochsson L, Gallagher AG, Hedman L, Hogman C, McClusky DA 3rd, Ramel S, Smith CD, Arvidsson D. Proficiency-based virtual reality training significantly reduces the error rate for residents during their first 10 laparoscopic cholecystectomies. Am J Surg. 2007 Jun;193(6):797-804. doi: 10.1016/j.amjsurg.2006.06.050. PMID 17512301
- [Background] Gallagher AG, McClure N, McGuigan J, Ritchie K, Sheehy NP. An ergonomic analysis of the fulcrum effect in the acquisition of endoscopic skills. Endoscopy. 1998 Sep;30(7):617-20. doi: 10.1055/s-2007-1001366. PMID 9826140
- [Background] Crothers IR, Gallagher AG, McClure N, James DT, McGuigan J. Experienced laparoscopic surgeons are automated to the "fulcrum effect": an ergonomic demonstration. Endoscopy. 1999 Jun;31(5):365-9. doi: 10.1055/s-1999-26. PMID 10433045
- [Background] Ritter EM, McClusky DA 3rd, Gallagher AG, Enochsson L, Smith CD. Perceptual, visuospatial, and psychomotor abilities correlate with duration of training required on a virtual-reality flexible endoscopy simulator. Am J Surg. 2006 Sep;192(3):379-84. doi: 10.1016/j.amjsurg.2006.03.003. PMID 16920434
- [Background] Fried MP, Satava R, Weghorst S, Gallagher AG, Sasaki C, Ross D, Sinanan M, Uribe JI, Zeltsan M, Arora H, Cuellar H. Identifying and reducing errors with surgical simulation. Qual Saf Health Care. 2004 Oct;13 Suppl 1(Suppl 1):i19-26. doi: 10.1136/qhc.13.suppl_1.i19. PMID 15465950
- [Background] Gallagher AG, Ritter EM, Champion H, Higgins G, Fried MP, Moses G, Smith CD, Satava RM. Virtual reality simulation for the operating room: proficiency-based training as a paradigm shift in surgical skills training. Ann Surg. 2005 Feb;241(2):364-72. doi: 10.1097/01.sla.0000151982.85062.80. PMID 15650649
- [Background] Van Sickle KR, McClusky DA 3rd, Gallagher AG, Smith CD. Construct validation of the ProMIS simulator using a novel laparoscopic suturing task. Surg Endosc. 2005 Sep;19(9):1227-31. doi: 10.1007/s00464-004-8274-6. Epub 2005 Jul 21. PMID 16025195
- [Background] Delaney CP. Outcome of discharge within 24 to 72 hours after laparoscopic colorectal surgery. Dis Colon Rectum. 2008 Feb;51(2):181-5. doi: 10.1007/s10350-007-9126-y. Epub 2008 Jan 4. PMID 18175188
- [Background] Lordan JT, Tilney HS, Shirol S, Jourdan I, Gudgeon AM. Does the laparoscopic colorectal surgery learning curve adversely affect the results of colorectal cancer resection? A 3-year prospective study in a district general hospital. Colorectal Dis. 2008 May;10(4):363-9. doi: 10.1111/j.1463-1318.2007.01332.x. Epub 2007 Oct 19. PMID 17949448
- [Background] Ridgway PF, Boyle E, Keane FB, Neary P. Laparoscopic colectomy is cheaper than conventional open resection. Colorectal Dis. 2007 Nov;9(9):819-24. doi: 10.1111/j.1463-1318.2007.01221.x. Epub 2007 Mar 7. PMID 17477851
- [Background] Suzuki S, Eto K, Hattori A, Yanaga K, Suzuki N. Surgery simulation using patient-specific models for laparoscopic colectomy. Stud Health Technol Inform. 2007;125:464-6. PMID 17377327
- [Background] Hernandez JD, Bann SD, Munz Y, Moorthy K, Datta V, Martin S, Dosis A, Bello F, Darzi A, Rockall T. Qualitative and quantitative analysis of the learning curve of a simulated surgical task on the da Vinci system. Surg Endosc. 2004 Mar;18(3):372-8. doi: 10.1007/s00464-003-9047-3. Epub 2004 Feb 2. PMID 14752634
- [Background] Haque S, Srinivasan S. A meta-analysis of the training effectiveness of virtual reality surgical simulators. IEEE Trans Inf Technol Biomed. 2006 Jan;10(1):51-8. doi: 10.1109/titb.2005.855529. PMID 16445249
- [Background] Munz Y, Almoudaris AM, Moorthy K, Dosis A, Liddle AD, Darzi AW. Curriculum-based solo virtual reality training for laparoscopic intracorporeal knot tying: objective assessment of the transfer of skill from virtual reality to reality. Am J Surg. 2007 Jun;193(6):774-83. doi: 10.1016/j.amjsurg.2007.01.022. PMID 17512295
- [Background] Satava RM. Surgical education and surgical simulation. World J Surg. 2001 Nov;25(11):1484-9. doi: 10.1007/s00268-001-0134-0. PMID 11760753
- [Background] Seymour NE. Integrating simulation into a busy residency program. Minim Invasive Ther Allied Technol. 2005;14(4):280-6. doi: 10.1080/13645700500272421. PMID 16754176
- [Background] Aggarwal R, Ward J, Balasundaram I, Sains P, Athanasiou T, Darzi A. Proving the effectiveness of virtual reality simulation for training in laparoscopic surgery. Ann Surg. 2007 Nov;246(5):771-9. doi: 10.1097/SLA.0b013e3180f61b09. PMID 17968168
- [Background] Hedman L, Strom P, Andersson P, Kjellin A, Wredmark T, Fellander-Tsai L. High-level visual-spatial ability for novices correlates with performance in a visual-spatial complex surgical simulator task. Surg Endosc. 2006 Aug;20(8):1275-80. doi: 10.1007/s00464-005-0036-6. Epub 2006 Jul 24. PMID 16865624
- [Background] Boller AM, Nelson H. Colon and rectal cancer: laparoscopic or open? Clin Cancer Res. 2007 Nov 15;13(22 Pt 2):6894s-6s. doi: 10.1158/1078-0432.CCR-07-1138. PMID 18006796
- [Background] Delaney CP, Pokala N, Senagore AJ, Casillas S, Kiran RP, Brady KM, Fazio VW. Is laparoscopic colectomy applicable to patients with body mass index >30? A case-matched comparative study with open colectomy. Dis Colon Rectum. 2005 May;48(5):975-81. doi: 10.1007/s10350-004-0941-0. PMID 15793638
- [Background] Fleshman J, Sargent DJ, Green E, Anvari M, Stryker SJ, Beart RW Jr, Hellinger M, Flanagan R Jr, Peters W, Nelson H; Clinical Outcomes of Surgical Therapy Study Group. Laparoscopic colectomy for cancer is not inferior to open surgery based on 5-year data from the COST Study Group trial. Ann Surg. 2007 Oct;246(4):655-62; discussion 662-4. doi: 10.1097/SLA.0b013e318155a762. PMID 17893502
- [Background] Jayne DG, Guillou PJ, Thorpe H, Quirke P, Copeland J, Smith AM, Heath RM, Brown JM; UK MRC CLASICC Trial Group. Randomized trial of laparoscopic-assisted resection of colorectal carcinoma: 3-year results of the UK MRC CLASICC Trial Group. J Clin Oncol. 2007 Jul 20;25(21):3061-8. doi: 10.1200/JCO.2006.09.7758. PMID 17634484
- [Background] Bonjer HJ, Hop WC, Nelson H, Sargent DJ, Lacy AM, Castells A, Guillou PJ, Thorpe H, Brown J, Delgado S, Kuhrij E, Haglind E, Pahlman L; Transatlantic Laparoscopically Assisted vs Open Colectomy Trials Study Group. Laparoscopically assisted vs open colectomy for colon cancer: a meta-analysis. Arch Surg. 2007 Mar;142(3):298-303. doi: 10.1001/archsurg.142.3.298. PMID 17372057
- [Background] Daetwiler S, Guller U, Schob O, Adamina M. Early introduction of laparoscopic sigmoid colectomy during residency. Br J Surg. 2007 May;94(5):634-41. doi: 10.1002/bjs.5638. PMID 17330835
- [Background] Reza MM, Blasco JA, Andradas E, Cantero R, Mayol J. Systematic review of laparoscopic versus open surgery for colorectal cancer. Br J Surg. 2006 Aug;93(8):921-8. doi: 10.1002/bjs.5430. PMID 16845692
- [Background] Moore MJ, Bennett CL. The learning curve for laparoscopic cholecystectomy. The Southern Surgeons Club. Am J Surg. 1995 Jul;170(1):55-9. doi: 10.1016/s0002-9610(99)80252-9. PMID 7793496
- [Background] Haluck RS, Gallagher AG, Satava RM, Webster R, Bass TL, Miller CA. Reliability and validity of Endotower, a virtual reality trainer for angled endoscope navigation. Stud Health Technol Inform. 2002;85:179-84. PMID 15458082
- [Background] Satava RM. Virtual reality surgical simulator. The first steps. Surg Endosc. 1993 May-Jun;7(3):203-5. doi: 10.1007/BF00594110. PMID 8503081
- [Background] Taffinder N, Sutton C, Fishwick RJ, McManus IC, Darzi A. Validation of virtual reality to teach and assess psychomotor skills in laparoscopic surgery: results from randomised controlled studies using the MIST VR laparoscopic simulator. Stud Health Technol Inform. 1998;50:124-30. PMID 10180527
- [Background] Seymour NE, Gallagher AG, Roman SA, O'Brien MK, Bansal VK, Andersen DK, Satava RM. Virtual reality training improves operating room performance: results of a randomized, double-blinded study. Ann Surg. 2002 Oct;236(4):458-63; discussion 463-4. doi: 10.1097/00000658-200210000-00008. PMID 12368674
- [Background] Grantcharov TP, Kristiansen VB, Bendix J, Bardram L, Rosenberg J, Funch-Jensen P. Randomized clinical trial of virtual reality simulation for laparoscopic skills training. Br J Surg. 2004 Feb;91(2):146-50. doi: 10.1002/bjs.4407. PMID 14760660
- [Background] Dincler S, Koller MT, Steurer J, Bachmann LM, Christen D, Buchmann P. Multidimensional analysis of learning curves in laparoscopic sigmoid resection: eight-year results. Dis Colon Rectum. 2003 Oct;46(10):1371-8; discussion 1378-9. doi: 10.1007/s10350-004-6752-5. PMID 14530677
- [Background] Schlachta CM, Mamazza J, Seshadri PA, Cadeddu M, Gregoire R, Poulin EC. Defining a learning curve for laparoscopic colorectal resections. Dis Colon Rectum. 2001 Feb;44(2):217-22. doi: 10.1007/BF02234296. PMID 11227938
- [Background] Cowie R. Measurement and modelling of perceived slant in surfaces represented by freely viewed line drawings. Perception. 1998;27(5):505-40. doi: 10.1068/p270505. PMID 10070553
- [Background] Noldus LP, Trienes RJ, Hendriksen AH, Jansen H, Jansen RG. The Observer Video-Pro: new software for the collection, management, and presentation of time-structured data from videotapes and digital media files. Behav Res Methods Instrum Comput. 2000 Feb;32(1):197-206. doi: 10.3758/bf03200802. PMID 10758678